CLINICAL TRIAL: NCT00184756
Title: Effect of Two Years Treatment With Growth Hormone on Height in SGA Children.
Brief Title: Efficacy on Height in SGA Children Treated With Growth Hormone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHLIQUID-1424
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Europe and Middle East. Growth hormone in SGA Children This trial compares a treated group of patients with an untreated group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Born small for gestational age with length and/or weight at -2 SDS or below at time of birth, according to country specific references.
* Severe growth failure with no catch up and with height at -2.5 SDS or below, according to country specific references, for chronological age at time of inclusion

Exclusion Criteria:

* Growth Hormone Deficiency (GHD)
* Treatment with any medical product which may interfere with GH effects
* Growth retardation associated with infections, severe chronic diseases including chromosomal anomaly or nutritional disorders

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2002-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Evaluate effect on Height in SGA Children Treated with Growth Hormone | After 2 years of treatment

SECONDARY OUTCOMES:
Appetite
Height SDS, yearly

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (33):
- Czechia (4):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Usti N. Labem
- Finland (3):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
- Germany (5):
  - Novo Nordisk Investigational Site, Gotha
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Krefeld
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Wuppertal
- Israel (4):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rehovot
- Poland (3):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Warsaw
- Portugal (4):
  - Novo Nordisk Investigational Site, Coimbra
  - Novo Nordisk Investigational Site, Matosinhos Municipality
  - Novo Nordisk Investigational Site, Porto
  - Novo Nordisk Investigational Site, Vila Nova de Gaia
- Spain (7):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Esplugues Llobregat
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Valencia
- Sweden (3):
  - Novo Nordisk Investigational Site, Helsingborg
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Stockholm

REFERENCES:
- [Result] Phillip M, Lebl J, Zuckerman-Levin N, Korpal-Szczyrska M, Sales Marques J, Ibáñez L on behalf of the European Norditropin SGA study group. Multinational study in short SGA children: evaluation of the effect of three different growth hormone dose regimens. European Society for Paediatric Endocrinology (ESPE) 2007; Country: Finland City: Helsinki
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com